CLINICAL TRIAL: NCT00939068
Title: A Study of Efficacy and Safety of Telbivudine in Pregnancy for the Prevention of Perinatal Transmission of Hepatitis B Virus Infection
Brief Title: Efficacy and Safety Study of Telbivudine to Prevent Perinatal Transmission
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Southeast University, China (Other)
Responsible Party: Wei Zhao, the Second Hospital of Nanjing, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H200804
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Hepatitis B, Gestation
Keywords: Chronic hepatitis B, Telbivudine, Intrauterine transmission
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telbivudine (Experimental): Drug administration and follow up: the subjects in Telbivudine group start dosing Telbivudine orally at 20-32 gestational weeks, with 600 mg daily, continue to one month after delivery.And their newborns are given HBIG 200IU by injection immediately after born and at day 15. They are also injected with genetically engineered HB vaccine 20ug respectively at age of 0, 1 and 6 months.
  Interventions: Drug: Telbivudine
- Control (Other): The pregnant subjects in Control group are intervented with no drugs, but their newborns are given HBIG 200IU by injection immediately after born and at day 15. They are also injected with genetically engineered HB vaccine 20ug respectively at age of 0, 1 and 6 months.
  Interventions: Biological: engineered HB vaccine

INTERVENTIONS:
Drug: Telbivudine — Subjects start dosing Telbivudine orally at 20-32 gestational weeks, with 600 mg daily, continued to one month after delivery.
  Other Names: telbivudine treatment
  Arms: Telbivudine
Biological: engineered HB vaccine — All the newborns in control group are given HBIG 200IU by injection immediately after born and at day 15. They are also injected with genetically engineered HB vaccine 20 ug respectively at age of 0, 1 and 6 months.
  Other Names: control group
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Telbivudine in pregnancy for the prevention of HBV perinatal transmission in highly viraemic mothers.

DETAILED DESCRIPTION:
In the present study, we evaluated the effect of telbivudine given during the second and third trimesters of pregnancy to highly viremic, HBV DNA-positive mothers on maternal HBV DNA and HBeAg levels prior to delivery and the rate of vertical transmission of HBV to infants who received passive-active immunoprophylaxis. Additionally, we investigated the timing of the administration of telbivudine on reducing the risk of perinatal transmission and the safety of telbivudine during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years old pregnant woman with gestational age of 20-32 week;
* positive serum HBsAg;
* HBV DNA≥1.0x106 copies/ml;

Exclusion Criteria:

* with previous antiviral treatment;
* with clinical sign of threatened miscarriage or related treatment in early pregnancy;
* positive serum HAV, HCV, HDV and HEV tests;
* fetus deformity by 3-D ultrasound examination;
* on other dugs, such as immune modulators, cytotoxic drugs or steroids;
* husbands are infected with HBV.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-07 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
the intrauterine transmission rate;vertical transmission rate (intrauterine and delivery) | 1 month post partum

SECONDARY OUTCOMES:
liver function normalization rate; HBV DNA and HBeAg reduction and negative conversion rate; | 1 month post partum
drug adverse reaction in pregnant women; complications during pregnancy and delivery, gestational age at delivery, the method of delivery, peripartum hemorrhage, the newborn growth and development milestones, Apgar score, newborn deformity prevalence | .1 year after childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, P.H.D, Study Chair — the Second Affiliated Hospital of Southeast University

REFERENCES:
- [Derived] Han GR, Jiang HX, Wang CM, Ding Y, Wang GJ, Yue X, Zhou L, Zhao W. Long-term safety and efficacy of telbivudine in infants born to mothers treated during the second or third trimesters of pregnancy. J Viral Hepat. 2017 Jun;24(6):514-521. doi: 10.1111/jvh.12670. Epub 2017 Feb 14. PMID 28039902